CLINICAL TRIAL: NCT01878071
Title: The Effect of Obesity on Oral Peri-implant Health - A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: Osseointegration Foundation (Unknown); University of Iowa Institute of Clinical and Translational Science (Unknown)
Responsible Party: Sponsor
Other Study IDs: UIOB01
Record Dates: First submitted 2013-01-22; First posted 2013-06-14 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Obesity; Peri-implant Inflammation; Peri-implantitis
MeSH Terms: conditions — Obesity; Peri-Implantitis

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Single group cross sectional

SUMMARY:
In recent years, greater emphasis has been placed on the link between oral and systemic health. Obesity, a growing medical problem worldwide, has been associated with multiple chronic inflammatory diseases such as diabetes mellitus and cardiovascular disease. With respect to the effect of obesity on periodontal health, it has been shown that obese subjects exhibit higher inflammation around natural teeth and are at increased risk of tooth loss than individuals with normal weight. Peri-implantitis, an inflammatory condition of bacterial origin that occurs around oral implants and resembles periodontal disease, has become a serious concern for the dental profession given its increasing prevalence and challenging treatment. There is also strong evidence that individuals with a history of periodontitis are also at risk for peri-implantitis. However, knowledge about the pathogenesis and treatment of peri-implantitis is scarce. Hence, it is extremely important to understand the implications of excessive body fat on peri-implant health. Based on the current understanding on the effect of obesity on systemic and local inflammation around natural teeth, the investigators hypothesize that obesity will have a significant impact on peri-implant health by inducing an increased inflammatory response as measured by clinical as well as molecular markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Currently non-smokers
* Subjects in maintenance care with adequate dental plaque control (<20% plaque index according to O'Leary et al. 1972)
* Subjects with at least one rough surface titanium oral implant in function for at least 6 months.

Exclusion Criteria:

* Edentulous subjects or subjects presenting with blade-type implants and/or implants with smooth surface.
* Pregnant or nursing women
* Subjects who have taken medications that are known to alter the oral inflammatory status, such as antibiotics and anti-inflammatory agents, for 3 months prior to the study.
* Subjects with a history of aggressive periodontitis (As defined by the American Academy of Periodontology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in maintenance dental care with at least one rough surface titanium oral implant in function
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Degree of peri-implant inflammation | Single time point - during their single visit (day one)

CONTACTS AND LOCATIONS:
Locations (1):
- Craniofacial Clinical Research Center at the University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Koldsland OC, Scheie AA, Aass AM. Prevalence of peri-implantitis related to severity of the disease with different degrees of bone loss. J Periodontol. 2010 Feb;81(2):231-8. doi: 10.1902/jop.2009.090269. PMID 20151801
- [Background] Al-Zahrani MS, Bissada NF, Borawskit EA. Obesity and periodontal disease in young, middle-aged, and older adults. J Periodontol. 2003 May;74(5):610-5. doi: 10.1902/jop.2003.74.5.610. PMID 12816292